CLINICAL TRIAL: NCT01623388
Title: Epigenetic Modifications Induced by Glycemic Variability
Brief Title: Epigenetic Modifications of Diabetes Mellitus Type I
Status: Withdrawn | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute
Other Study IDs: 11-5649
Record Dates: First submitted 2012-06-07; First posted 2012-06-20 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Type I Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucose Tolerance Test; Clinical Trials, Phase I as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood

GROUPS / COHORTS (1):
- Phase I
  Interventions: Procedure: Oral glucose tolerance test for Phase I

INTERVENTIONS:
Procedure: Oral glucose tolerance test for Phase I — Oral glucose tolerance test for Diabetic patients in phase I

SUMMARY:
This research is being done to find out if significant changes in blood glucose cause bad outcomes in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Diagnosis of Type I diabetes
* Willing to wear continuous blood glucose monitor as specified in protocol

Exclusion Criteria:

* Pregnant or planning to become pregnant during the study

Healthy control group Inclusion:

* 18-65 years old
* Willing to wear continuous blood glucose monitor as specified in protocol

Exclusion:

* Pregnant or planning to become pregnant during the study
* Diagnosis of Type I or II Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type I Diabetic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Evaluate blood sugar variability in Type I diabetics for differences in epigenetic signatures between Type I diabetics with little glycemic variability as compared to those with more pronounced glycemic changes. | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps, San Diego, California, United States